CLINICAL TRIAL: NCT06430593
Title: Evaluation of Low Flow and Normal Flow Anesthesia Management in Robotic Assisted Laparoscopic Surgeries
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Hilal AKCA, Anesthesiologist, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024- 183
Record Dates: First submitted 2024-05-14; First posted 2024-05-28 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-05

CONDITIONS: Oncology
Keywords: low-flow anesthesia; robotic-assisted surgery; general anesthesia
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low-flow anesthesia: 0,5 lt/min
  Interventions: Procedure: low-flow anesthesia
- normal flow anesthesia: >1 lt/min
  Interventions: Procedure: low-flow anesthesia

INTERVENTIONS:
Procedure: low-flow anesthesia — 0,5 l/min >1 l/min
  Other Names: normal flow anesthesia

SUMMARY:
Robotic-assisted laparoscopic surgery has many advantages compared to conventional open surgery, such as less postoperative pain, shorter hospital stays, and faster recovery times. Robot-assisted surgeries require general anesthesia. In our clinic, we routinely apply low-flow anesthesia methods in addition to normal flow methods in many surgical applications, according to clinician preferences. The aim of this study is to determine the effects of low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia applications in robotic-assisted laparoscopic surgeries.

To compare perioperative hemodynamic and respiratory parameters in terms of inhalation agent and soda lime consumption.

DETAILED DESCRIPTION:
Robotic surgery is the performance of laparoscopic surgery using a robotic interface. The robotic surgery system used today is called Da Vinci S. In surgeries performed with the help of a robot, the surgeon can work more precisely and with greater maneuverability. Therefore, an operation can be performed that is less traumatic for the patient than other methods.Robotic-assisted laparoscopic surgery has many advantages compared to conventional open surgery, such as less postoperative pain, shorter hospital stays, and faster recovery times. Robot-assisted surgeries require general anesthesia. In these applications, fresh gas flow in anesthesia systems can be made with traditional high, normal or low flow strategies, depending on the preference of the clinicians.Low-flow anesthesia creates a breathing air closer to physiological conditions during anesthesia by heating and humidifying the inhaled gases. In addition, it provides cost advantage by reducing inhalation agent consumption and reduces atmospheric pollution. It is suggested that the use of both fresh gas flow amounts does not pose a safety risk for patients, and that the use of low-flow anesthesia methods should be more widespread due to the advantages it provides. In our clinic, investigators routinely apply low-flow anesthesia methods in addition to normal flow methods in many surgical applications, according to clinician preferences. The aim of this study is to determine the effects of low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia applications in robotic-assisted laparoscopic surgeries.

To compare perioperative hemodynamic and respiratory parameters in terms of inhalation agent and soda lime consumption.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* ASA I,II
* Patients undergoing robotic-assisted laparoscopic surgery

Exclusion Criteria:

* ASA III,IV,V
* Those with serious cardiac, respiratory, hepatic, renal disease
* People with mental status disorders, psychiatric illnesses
* Patients with hearing problems and glaucoma
* Desire to be out of work

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ages 18-75, ASA I,II, Patients undergoing robotic-assisted laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Parameters | Perioperative period(approximately 3-6 hours)
  It was aimed to compare heart rates in patients undergoing low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia.
Hemodynamic Parameters | Perioperative period(approximately 3-6 hours)
  It was aimed to compare blood pressure in patients undergoing low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia.
Respiratory parameters | Perioperative period(approximately 3-6 hours)
  It was aimed to compare oxygen saturation in patients undergoing low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia.
Respiratory parameters | Perioperative period(approximately 3-6 hours)
  It was aimed to compare endtidal carbon dioxide in patients undergoing low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia.
Inhalation agent (sevoflurane) consumption | Perioperative period(approximately 3-6 hours)
  It was aimed to compare inhalation agent (sevoflurane) consumption (lt) in patients undergoing low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia.
Soda lime consumption | Perioperative period(approximately 3-6 hours)
  It was aimed to compare soda lime consumption in patients undergoing low flow (0.5 lt/min) and normal flow (>1 lt/min) anesthesia.
  Soda lime consumption refers to the number of changes of the soda lime canister.